CLINICAL TRIAL: NCT06934616
Title: A Phase I, First-in-Human, Open-Label, Multicenter Study Evaluating the Safety, Tolerability, Pharmacokinetics and Efficacy of a Trispecific PD-1/CTLA-4/ VEGF Antibody GB268 in Participants With Advanced Solid Tumors
Brief Title: A Phase I, First-in-Human Study of GB268 (PD-1/CTLA-4/VEGF Trispecific Antibody) in Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GB268-001
Record Dates: First submitted 2025-03-16; First posted 2025-04-18 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor Cancer
Keywords: PD-1; CTLA-4; VEGF; anti-PD-1/CTLA-4/VEGF trispecific antibody; advanced solid tumors; Phase I
MeSH Terms: conditions — Diabetes Mellitus, Insulin-Dependent, 12

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GB268 (Experimental)
  Interventions: Drug: GB268

INTERVENTIONS:
Drug: GB268 — GB268 will be administered via intravenous infusion once every 3 weeks on Days 1 of each 21-day cycle

SUMMARY:
This is a Phase I, First-in-Human, Open-Label, Multicenter Study Evaluating the Safety, Tolerability, Pharmacokinetics and Efficacy of a Trispecific PD-1/CTLA-4/VEGF Antibody GB268 in Participants with Advanced Solid Tumors. The study will consist of a dose-escalation stage and an dose-expansion stage.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of Informed Consent.
2. Able to give voluntary informed consent and are willing to follow and complete all the study required procedures.
3. Participants with histologically or cytologically confirmed locally advanced, metastatic or unresectable solid tumors that have failed standard therapy, or for whom no standard therapy exists, or where standard therapy is contraindicated.
4. Participants must have measurable disease according to Response Criteria in Solid Tumors (RECIST) v1.1.
5. ECOG performance status ≤ 1.
6. Participants with HCC must have a Child-Pugh score class A.
7. Life expectancy ≥ 3 months.
8. Participants must have adequate organ function
9. Tumor tissue samples for biomarker testing are highly desirable (mandatory in dose expansion part)
10. For women of childbearing potential: participants must have a negative serum pregnancy test within 7 days prior to Cycle 1 Day 1 and agree to abstain from heterosexual intercourse or use an acceptable contraceptive method during the study and for at least 6 months following the final administration of GB268.
11. For male participants: agreement to abstain from heterosexual intercourse or use of an acceptable contraceptive method during the study treatment and for at least 6 months following the final infusion, and agreement to refrain from sperm donation during the study treatment and for at least 6 months following the final administration of GB268.

Exclusion Criteria:

1. Received the following treatments or medications before starting the study treatment:

   1. Participants who received the last systemic anti-tumor therapy, including chemotherapy, biological agents etc., within 3 weeks prior to Cycle 1 Day 1; participants who received hormonal anti-tumor therapy and small molecule targeted therapy within 2 weeks prior to Cycle 1 Day 1; and participants who received Chinese herbal medicine or traditional Chinese medicinal products with anti-tumor indications within 2 weeks prior to Cycle 1 Day 1. Participants who received non-specific immunomodulatory therapy (e.g., interleukin, interferon, thymosin, tumor necrosis factor, etc.) within 2 weeks prior to Cycle 1 Day 1.
   2. Received a live or attenuated vaccination within 4 weeks prior to Cycle 1 Day 1.
   3. Prior radiation therapy completed within 3 weeks prior to Cycle 1 Day 1. Palliative radiotherapy for the control of symptoms is allowed to be completed at least 2 weeks prior to Cycle 1 Day 1.
2. Treatment with systemic immunosuppressive medications within 2 weeks prior to Cycle 1 Day 1.
3. Participants who have, or will have, any of the following:

   1. An invasive operative procedure within 4 weeks of, or with incomplete recovery, before Cycle 1 Day 1. Participants who have undergone minor local procedure (excluding peripherally inserted central catheterisation and intravenous infusion port implantation) within 3 days prior to Cycle 1 Day 1.
   2. Significant traumatic injury within 4 weeks prior to Cycle 1 Day 1 (all wounds must be fully healed prior to Cycle 1 Day 1).
   3. Any medical condition that affects wound healing capacity and is expected to endanger participant safety if wound healing capacity would be severely reduced during administration of the investigational product.
   4. Major surgery expected during study participation.
4. Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Grade ≤ 1
5. Participants who have experienced ≥ Grade 3 immune-related adverse events (irAE) or irAE leading to treatment discontinuation
6. Has known active central nervous system (CNS) metastases.
7. Participants with a history of other malignancies unless the patient has undergone potentially curative therapy with no evidence of that disease for 3 years prior to Cycle 1 Day 1
8. Uncontrolled pleural effusion, or ascites requiring recurrent drainage procedures within 4 weeks prior to Cycle 1 Day 1.
9. History of clinically significant cardiovascular disease.
10. History of interstitial lung disease (ILD).
11. Active or prior documented autoimmune disease required systemic treatment within the past 2 years.
12. Active or prior history of inflammatory bowel disease (such as Crohn's disease, ulcerative colitis, or chronic diarrhea).
13. Prior history of hypertensive crisis or hypertensive encephalopathy.
14. Participants with significant coagulation disorders or other obvious evidence of bleeding risk.
15. History of abdominal fistula, tracheoesophageal fistula, and female genital fistula (e.g., vesicovaginal fistula, urethrovaginal fistula, and vesicocervical fistula, etc.), gastrointestinal perforation, or abdominal abscess, or patient has risk factors for gastrointestinal obstruction at the discretion of the investigator.
16. Active infection that have received systemic anti-infective treatment within 2 weeks prior to Cycle 1 Day 1. Serious infections within 4 weeks prior to Cycle 1 Day 1, including but not limited to complications requiring hospitalization, sepsis or severe pneumonia.
17. Participants with uncontrolled concurrent illness, including, but not limited to, poorly controlled hypertension or Type 2 diabetes mellitus, or psychiatric illness or a social situation that would limit compliance with the study requirements.
18. Known presence of active tuberculosis.
19. Participants have at screening:

    1. Positive hepatitis B (hepatitis B virus [HBV]) surface antigen (HBsAg) or Hepatitis B Core Antibody (HBcAb), with HBV-DNA result greater than 500 IU/mL (or 2500 copies/mL).
    2. Positive hepatitis C virus antibody (anti-HCV), with HCV-RNA result greater than the lower limit of quantification.
20. History of primary immunodeficiency. Participants who have previously been positive for human immunodeficiency virus (HIV) antibody, or are positive for HIV at screening.
21. History of solid organ or blood system transplantation, except for corneal transplantation.
22. Female patients who are pregnant, or breast-feeding.
23. Patients with known allergies, hypersensitivity, or intolerance to GB268 or its excipients. Patients with history of severe hypersensitivity reactions to other mAbs.
24. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2025-04-24 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to approximately 2 years
  Safety as assessed by clinical laboratory tests, 12-lead electrocardiogram (ECG), vital signs measurements, and the incidence, nature and severity of all adverse events (AEs) and serious AEs (SAEs)
Dose Limiting Toxicity (DLT) | 21 days
  Incidence of Dose Limiting Toxicity (DLT) during the first cycle of treatment

SECONDARY OUTCOMES:
ORR | Up to approximately 2 years
  objective response rate assessed by investigator per RECIST v1.1
DOR | Up to approximately 2 years
  duration of response assessed by investigator per RECIST v1.1
DCR | Up to approximately 2 years
  disease control Rate assessed by investigator per RECIST v1.1
PFS | Up to approximately 2 years
  progression free survival assessed by investigator per RECIST v1.1
Cmax of GB268 | Up to approximately 2 years
  Peak plasma concentration
Tmax of GB268 | Up to approximately 2 years
  Time to peak drug concentration
AUC of GB268 | Up to approximately 2 years
  Area under curve
ADA of GB268 | Up to approximately 2 years
  Detection of anti-GB268 antibodies

IPD SHARING:
Plan to Share IPD: No